CLINICAL TRIAL: NCT04625452
Title: Feasibility and Efficacy of Lifestyle Risk Factors Through Brief Behaviour Change Counseling in NCD's Participants Using 5A's and a Guiding Style (BBCC+ 5A's +GS) in Mangochi, Southern Malawi
Brief Title: Feasibility and Efficacy of Brief Behavior Change Counseling on Lifestyle in Hypertensive and Diabetics Participants
Acronym: BBCC+5A's+GS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kamuzu University of Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P.08/18/2454; 5U24HL136791-01 (NIH)
Record Dates: First submitted 2020-08-19; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Hypertension; Diabetes; Life Style
Keywords: lifestyle; diabetics; hypertensives; brief behavior change; counseling; motivational interviewing; 5 A's
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Intervention group will be administered at 3, 12 and 24 weeks. The intervention consists in addition to normal care and distribution of printed education pamphlets, of an individual counseling based on lifestyle risk factors of diabetic or hypertensive participants themed around 5 points (ask, advice or alert, assess , assist and arrange). It will use a guiding style from motivational interviewing consisting of asking opened questions, summarizing patients, reflecting him his statements, and capture change words, and requesting for permission to introduce any new point.
  Normal care Participants allocated to normal care (control group) will receive standard care for diabetes or hypertension as per Malawi- government's NCD's guidelines: drugs, inconsistent unstructured advises regarding lifestyle behavior, opportunistic biological tests as per clinician's judgement.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The data will be collected under investigator's supervision, documented by nurses ( counselors), clinical officers ( doing routine consultations), lab technicians ( analyzing blood) and the clerk doing the measurements. Data sent to the investigators and statisticians for entry and analysis will be blinded beforehand by removing the identifiers' information. After completing the analysis, results will be again allocated to their respective arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BBCC+5A's+GS (Experimental): Brief behavior change counseling using 5A's + Guiding style (from motivational interviewing) + Printed education materials ( at baseline, 12 weeks, 24 weeks)
  Interventions: Behavioral: BBCC+5A's+GS
- Normal care (No Intervention): They will receive the normal care: simple advice on changing lifestyle risk factors + medications for diabetes or hypertension ( at baseline, 12 weeks, 24 weeks)

INTERVENTIONS:
Behavioral: BBCC+5A's+GS — It is a 5-steps intervention delivered in a motivational interviewing spirit. Clearly the five steps are asking about the behaviour risk factors, assessing the level of risk factors; providing information about the pros and cons of the behaviour in a neutral way; assessing the change by probing about the importance in and the confidence of changing the risk factor; assisting the patient to come-up with a road map about changing the risk factor, connecting the patient to support networks or drugs which can increase the likelihood to change; and arranging for the next visit.
  All this given by asking opened question to participant, active listening, summarizing what he is saying, evoking change through concepts or statements, empathy and asking permission to provide further information.
  Other Names: Brief behavior change using 5A's and a guiding style from motivational interviewing
  Arms: BBCC+5A's+GS

SUMMARY:
The purpose of this study will be to assess the feasibility and the preliminary efficacy of brief behavior change counseling on lifestyle among diabetic and hypertensive patients

DETAILED DESCRIPTION:
1. BACKGROUND Noncommunicables diseases (NCDs) are on the rise globally as well as in Malawi, alongside their behavioral modifiable risk factors. Behavioral intervention such as brief behavior change counseling using 5A's and a guiding style (BBCC + 5As +GS) has shown an effect on reducing these lifestyles risk factors. Their effectiveness varies between the behavioral technique used. But So far, available evidences of this effect are from western countries. Even implementation of these techniques has been done in some countries, but so far there is no information about their implementation in noncommunicable diseases field in Mangochi, even Malawi. Therefore, a really need to conduct this study in Mangochi, Southern Malawi.
2. OBJECTIVES

   1. Overall objective: The primary objective of the study is to test the feasibility of the brief behavior change counseling using 5 A's and a guiding style from motivational interviewing which will be used for NCDs 'patients and assess its efficacy in improving lifestyle risk factors in NCDs' patients.
   2. Specific objectives for this study are

1. to evaluate the feasibility of participating in a future quasi-experimental study of BBCC + 5A's + GS ; 2. to estimate the efficacy of BBCC + 5A's + GS from MI on lifestyle risk factors, theory constructs, quality of life domains; 3. to provide data on which to estimate the sample size required to detect a statistically significant difference between experimental and control groups; 4. and to explore experience of participants and care providers during the brief behaviour change counseling sessions to NCDs' patients in Mangochi

4. Methodology:

1. Design: mixed methods (pilot quasi-experimental and qualitative study)
2. Settings: The study will take place at two sites: Mangochi District Hospital and Monkey Bay Community Hospital; Malawi.
3. sample size: Purposeful sampling and successive eligible patients. Sample size: Efficacy study will be conducted on 50 patients.
4. Intervention: brief behaviour change using 5A's and a Guiding style from motivational interviewing will be administered to participants in the intervention group by trained counsellors (nurses).

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-65 years old,
* registered in the clinic at least for 6 months,
* been screened for at least 1 lifestyle risk factor,
* express willingness to participate in the study,
* being permanent resident in Mangochi District for at least 12 months from recruitment, and
* Fluent in Chichewa and/or Yao

Exclusion Criteria:

* - present with any concomitant severe disease,
* being pregnant
* patient with an active Psychiatrics' comorbidity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-02-23 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
A measure of participants recruited (recruitment rate) | [Time frame: through study completion, an average of 24 weeks]
  The number of individuals recruited from those eligible
Number participants who consented to take part in the study | [Time frame: through study completion, an average of 24 weeks]
  The number of participants who accepted to take part in the study from those deemed eligible for the study
Proportion of participants who completed the study during the 12 weeks' period | [ time frame: up to 12 weeks]
  The number of participants who were able to complete each PROM divided by the total number of participants at 12 weeks
Proportion of participants who completed the study during the 24 weeks' period | [ Time frame: through study completion, an average of 24 weeks]
  The number of participants who were able to complete each PROM divided by the total number of participants at 24 weeks
Proportion of participants retained in the study | [ Time frame: through study completion, an average of 24 weeks]
  Proportion of participants who remained in the study during its full duration. The number of participants who are in the study at 6 months divided by the total number of patients who were recruited
Proportions of participant's loss-to-follow-up at 12 weeks | [ time frame: up to 12 weeks]
  Participants who stop (withdraw/dropout) and did not attend the 12 weeks' follow-up visit by the total of recruited participants.
Loss-to-follow-up at 24 weeks | [ Time frame: through study completion, an average of 24 weeks]
  Participants who stop (withdraw/dropout) and did not attend the 24 weeks' follow-up visit

SECONDARY OUTCOMES:
Change from baseline in Alcohol Use Disorder Identification Test-C at 12 weeks | [ Time frame: at baseline and in 12 weeks]
  Audit-C is a validated, self-reported measure of perceived severity (quantity and frequency) of consumption of alcohol comprising 3 questions whose score gives a global score from the 3.
  The scoring system of AUDIT-C is as follow: frequency of drink containing alcohol (scores: 0-4); number of standard drinks on a day (scores: 0-4); and frequency of 5 or more standard drinks on any one occasion (scores: 0-4). This global score is either below 5 (non-harmful alcohol use), or from 5 and higher (harmful alcohol). The higher the score, the severe the drinking.
Alcohol Use Disorder Identification Test-C at 24 weeks | [ Time frame: through study completion, an average of 24 weeks]
  Mean change from baseline of Alcohol Use Disorder Identification Test among participants who were screened for harmful alcohol use with a score of 5 or more on AUDIT-C at 24 weeks. 9. Change from baseline in Alcohol Use Disorder Identification Test-C at 12 weeks Audit-C is a validated, self-reported measure of perceived severity (quantity and frequency) of consumption of alcohol comprising 3 questions whose score gives a global score from the 3.
  The scoring system of AUDIT-C is as follow: frequency of drink containing alcohol (scores: 0-4); number of standard drinks on a day (scores: 0-4); and frequency of 5 or more standard drinks on any one occasion (scores: 0-4). This global score is either below 5 (non-harmful alcohol use), or from 5 and higher (harmful alcohol). The higher the score, the severe the drinking.
Mean change in smoking from baseline to 12 weeks using Short Fagerström Test for Nicotine dependence among participants who are screened for smoking of any form (cigarettes, chewing, tobacco, pipe) and any amount out at 24 weeks | [ Time frame: at baseline and 24 weeks]
  Fagertrom test using two questions for scoring related to time between walking-up and taking the first cigarettes (≤ 5 min= 3, 6-30 minutes=1, 31-60 minutes=3), and number of cigarettes taken per day (≤ 10=0, 11-20=1, 21-30=2, and ≥ 31=3). score varies from 0-6; 0-3=very low risk and 6= very high risk
Mean change in smoking from 12 weeks to 24 weeks using Short Fagerström Test for Nicotine dependence | [ Time frame: at 12 weeks and 24 weeks]
  Mean change in smoking from baseline to 12 weeks using Short Fagerström Test for Nicotine dependence among participants who are screened for smoking of any form (cigarettes, chewing, tobacco, pipe) and any amount out at 24 weeks. Fagertrom test using two questions for scoring related to time between walking-up and taking the first cigarettes (≤ 5 min= 3, 6-30 minutes=1, 31-60 minutes=3), and number of cigarettes taken per day ( ≤ 10=0, 11-20=1, 21-30=2, and ≥ 31=3). score varies from 0-6; 0-3=very low risk and 6= ery high risk
16. Change from 12 weeks in health-related quality of life using the World Health Organization quality of life tool (WHOQOL-Bref) | [Timeframe baseline, 12 weeks]
  WHOQoL-Bref is a validated, self-reported instrument that is a general measure of perceived health status comprising 26 questions and yielding to 5 scores from 5 dimensions (with subscales) that assess 5 dimensions, namely: mobility; self-care; usual activities; pain/discomfort; and anxiety/ depression. Each dimension has 3 levels: no problems, some problems, and extreme problems, with scores of 1, 2, and 3 representing each level, respectively. The Global score is given by the sum of scores in each dimension/domain. The change will be the differences in scores between the figures at 24 weeks' menus figures at 12 weeks. The low the score, the worse the quality of life.
  Score is given by the sum of scores in each dimension/domain. The change will be the differences in scores between the figures at 12 weeks' menus figures at baseline. The low the score, the worse the quality of life.
Change from baseline in health-related quality of life using the World Health Organization quality of life tool (WHOQOL-Bref) | [Timeframe: baseline and in 6 weeks]
  WHOQoL is a validated, self-reported instrument that is a general measure of perceived health status comprising 26 questions and yielding to 5 scores from 5 dimensions (with subscales) that assess 5 dimensions, namely: mobility; self-care; usual activities; pain/discomfort; and anxiety/ depression. Each dimension has 3 levels: no problems, some problems, and extreme problems, with scores of 1, 2, and 3 representing each level, respectively.
  The Global score is given by the sum of scores in each dimension/domain. The change will be the differences in scores between the figures at 12 weeks' menus figures at baseline. The low the score, the worse the quality of life.
Change in theory of planned behavior constructs' scores from baseline to 12 weeks | [Timeframe: baseline, 12 weeks]
  18. Change in theory of planned behavior constructs' scores from baseline to 12 weeks The theory of planned behavior posits that he fact for someone to perform a given behavior (example: adopts a healthy diet) is guided by three kinds of considerations: beliefs about the likely consequences and experiences associated with the behavior (behavioral beliefs), beliefs about the normative expectations and behaviors of significant others (normative beliefs), and beliefs about the presence of factors that may facilitate or impede performance of the behavior (control beliefs). To measure those three components, a 7 points-scale was applied to each behavior with high number representing better (positive numbers)/worse outcomes (negative numbers). For attitude: bad-good; pleasant-unpleasant For perceived norm (agree-disagree; unlikely-likely), for perceived behavioral control (true-false, disagree-agree); intension (likely-unlikely, false-true) . The higher the score, the better
Change in theory of planned behavior constructs' means' difference from 12 to 24 weeks | [Timeframe: 12 weeks through 24 weeks]
  The theory of planned behavior posits that he fact for someone to perform a given behavior (example: adopts a healthy diet) is guided by three kinds of considerations: beliefs about the likely consequences and experiences associated with the behavior (behavioral beliefs), beliefs about the normative expectations and behaviors of significant others (normative beliefs), and beliefs about the presence of factors that may facilitate or impede performance of the behavior (control beliefs).
  To measure those components, a 7 points-scale was applied to each behavior with high number representing better (positive numbers)/worse outcomes (negative numbers).
  Descriptive statistics per constructs were calculated. For attitude: bad-good; pleasant-unpleasant; for perceived norm (agree-disagree; unlikely-likely); for perceived behavioral control (true-false, disagree-agree); and intension (likely-unlikely, false-true)
To assess the change of the the theory of planned behavior constructs between baseline scores and 24 weeks' | [Time frame: 12, 24 weeks]
  The theory of planned behavior posits that he fact for someone to perform a given behavior (example: adopts a healthy diet) is guided by three kinds of considerations: beliefs about the likely consequences and experiences associated with the behavior (behavioral beliefs), beliefs about the normative expectations and behaviors of significant others (normative beliefs), and beliefs about the presence of factors that may facilitate or impede performance of the behavior (control beliefs).
  To measure those components, a 7 points-scale was applied to each behavior with high number representing better (positive numbers)/worse outcomes (negative numbers).
  Descriptive statistics per constructs were calculated. For attitude: bad-good; pleasant-unpleasant; for perceived norm (agree-disagree; unlikely-likely); for perceived behavioral control (true-false, disagree-agree); and intension (likely-unlikely, false-true)
Change of Trans theoretical model (TTM) stage from baseline to 12 weeks in the "Theoretical Model of Change" score | [time frame: baseline, 12 weeks]
  Change of Trans theoretical model (TTM) stage from baseline to 12 weeks in the "Theoretical Model of Change" score TTM is a validated, self-report tool used to detect the level of change a participant has at a given time. For our case at baseline, 12 weeks, and at 24 weeks) scored from 1 to 5. Comparison of the scoring at 12 and at 24 will show if there has been change or not.
  The staging system of TTM is as follow
  1. STAGE 1; pre contemplation: I do not intend in the next 6 months
  2. stage 2. Contemplation: I intend to in the next 6 months
  3. stage 3. Preparation: I intend to in the next 30 days
  4. stage 4. Action: have been doing so for less than 6 months
  5. stage 5 maintenance I have been doing so for more than 6 months The higher the stage, the advanced the degree of changes and vice-versa. Same figure at two different time points= no progress on degree of behavior change.
Change of TTT sub-scales means from 12 to 24 weeks in the "Theoretical Model of Change" scores | [Time frame: 12 weeks and 24 weeks]
  Change of Trans theoretical model (TTM) stage from baseline to 12 weeks in the "Theoretical Model of Change" score TTM is a validated, self-report tool used to detect the level of change a participant has at a given time. For our case at baseline, 12 weeks, and at 24 weeks) scored from 1 to 5. Comparison of the scoring at 12 and at 24 will show if there has been change or not.
  The staging system of TTM is as follow
  1. STAGE 1; pre contemplation: I do not intend in the next 6 months
  2. stage 2. Contemplation: I intend to in the next 6 months
  3. stage 3. Preparation: I intend to in the next 30 days
  4. stage 4. Action: have been doing so for less than 6 months
  5. stage 5 maintenance I have been doing so for more than 6 months The higher the stage, the advanced the degree of changes and vice-versa. Same figure at two different time points= no progress on degree of behavior change.

OTHER OUTCOMES:
change from baseline in body weight at 12 weeks | [Time frame: baseline and 12 weeks]
  The measure will be assessed in the morning before the clinic, participants will be weighted in light clothes, barefoot using bathroom scale and will be recorded to the nearest 0.1 kg. Change will be calculated as the difference of weight recorded at baseline and weight recorded at 12 weeks.
Change of body weight from 12 weeks at 24 weeks | [Time frame 12 and 24 weeks]
  The measure will be assessed in the morning before the clinic, participants will be weighted in light clothes, barefoot using bathroom scale and will be recorded to the nearest 0.1 kg. Change will be the difference of weight recorded at 12 weeks and weight recorded at 24 weeks.
Mean's change from baseline in Body Mass Index at 12 weeks | [Time Line: baseline and 12 weeks]
  The measure will be assessed after measurements of weight (kilograms) and height (meters) by dividing the weight square by the root-square of height (in meters). The values of below 18.5= underweight, 18.5-25= healthy weight, 25-29.9= overweight, and 30-35 = Grade I, 35-40: Grade II.,, ≥ 40: Grade III. Change will be the difference of BMI calculated at baseline and at 12 weeks. The higher the figure after 25, the worse the outcome.
Mean's Change from 12 weeks in Body Mass Index to 24 weeks | [Time Line: 12 weeks and 24 weeks]
  The measure will be assessed after measurements of weight (kilograms) and height (meters) by dividing the weight square by the root-square of height (in meters). The values of below 18.5= underweight, 18.5-25= healthy weight, 25-29.9= overweight, and 30-35 = Grade I, 35-40: Grade II.,, ≥ 40: Grade III.
  Change will be the difference of BMI calculated at 12 weeks with the figure at 24 weeks. The higher the figure after 25, the worse the outcome. The higher the figure after 25, the worse the outcome
Means' Change from baseline in Body Mass Index to 24 weeks | [Time Frame: baseline and 24 weeks]
  The measure will be assessed after measurements of weight (kilograms) and height (meters) by dividing the weight square by the root-square of height (in meters). The values of below 18.5= underweight, 18.5-25= healthy weight, 25-29.9= overweight, and 30-35 = Grade I, 35-40: Grade II.,, ≥ 40: Grade III. Change will be the difference of BMI calculated at baseline with the figure at 24 weeks. The higher the figure after 25, the worse the outcome
Means' Change in waist -to- hip ratio at 12 weeks | [Time Line: baseline and 12 weeks]
  Hip measurements were taken using a tape-measure placed horizontally at the point of maximum circumference over the buttocks. Measurements were taken to the nearest 0.1 cm.
Mean's change in Mean waist-to-hip ratio (WHR) at 12 weeks | [ Time Frame: baseline and 12 weeks]
  The measure will be assessed by dividing the waist circumference (using a tape-measure placed horizontally at the point between the iliac crest process and the lower margin of the last palpable rib in a patient standing on deep respiratory) by the hip circumference (Hip measurements were taken using a tape-measure placed horizontally at the point of maximum circumference over the buttocks) on a standing-up participants in deep expiration.
  The normal range value is 0.80- 0.75. High values Change will be the difference of WHR calculated at baseline with the figure at 24 weeks.
Mean's change in Mean waist-to-hip ratio at 24 weeks | [ Time Frame: baseline and 24 weeks]
  The measure will be assessed by dividing the waist circumference (using a tape-measure placed horizontally at the point between the iliac crest process and the lower margin of the last palpable last rib in a patient standing on deep respiratory) by the hip circumference (Hip measurements were taken using a tape-measure placed horizontally at the point of maximum circumference over the buttocks) on a standing-up participants in deep expiration.
  The normal range value from 0.80 to 0.70 More than……… central obesity. Change will be the difference of WRH calculated at 12 weeks and that at 24 weeks.
Means' Change from baseline in pulse rate using an electronic blood pressure machine | [Time frame: baseline and 12 weeks]
  This measure was assessed in the morning before the clinic alongside with the blood pressure recording through an electronic machine which is recording concurrently the blood pressure reading and the pulse rate. The normal values vary between 60-100, beyond which we have a tachycardia in adults, and below we note a bradycardia.
  The value change was calculated as the value recorded at baseline minus the value recorded before any clinical examination at 12 weeks.
Means' change from 12 weeks in pulse rate using an electronic blood pressure machine | [Time frame: 12 and 24 weeks]
  This measure was assessed in the morning in patient relaxed in seating position before the clinic alongside with the blood pressure. The third recorded pulse rate's reading from the battery powered digital blood pressure machine was recorded. The normal values varied between 60-100, beyond which we have a tachycardia in adults, and below we note a bradycardia.
  The value change was calculated as the value recorded at 12 weeks minus the value recorded at 24 weeks.
34. Means' change from baseline in the mean pulse rate to 24 weeks using an electronic blood pressure machine | [Time frame: baseline and 24 weeks]
  This measure was assessed in the morning before the clinic alongside with the blood pressure. The third recorded pulse rate's reading from the battery powered digital blood pressure machine was recorded. The normal values vary between 60-100, beyond which we have a tachycardia in adults, and below we note a bradycardia.
  The value change was calculated as the value recorded at baseline minus the value recorded before at 24 weeks.
35. Means' Change from baseline in the seated through cuff mean systolic blood pressure (SBP) from baseline to 12 weeks | [Time Frame: baseline and 12 weeks]
  The difference of the mean of third and second recorded systolic blood pressure readings on a seated relaxed patient from the battery powered digital blood pressure machine was recorded.
Mean's change from 12 weeks in the seated patient through cuff mean systolic blood pressure from 12 to 24 weeks | [Time Frame: 12 weeks and 24 weeks]
  The difference of the means of third and second recorded systolic blood pressure readings of the 12 and 24 weeks on a seated relaxed patient from the battery powered digital blood pressure machine was recorded.
Mean's change from baseline in the seated through cuff mean systolic blood pressure (SBP) from baseline to 12 weeks | [Time Frame: baseline and 12 weeks]
  The difference of the mean of third and second recorded systolic blood pressure readings on a seated relaxed patient from the battery powered digital blood pressure machine was recorded.
Mean's change from baseline in the seated patient through cuff mean systolic blood pressure from 0 to 24 weeks | [Time Frame: baseline and 24 weeks]
  The difference of the means of third and second recorded systolic blood pressure readings of the 0 and 24 weeks on a seated relaxed patient from the battery powered digital blood pressure machine was recorded.
Mean's change from baseline in the seated through cuff mean diastolic blood pressure (SBP) from baseline to 12 weeks | [Time Frame: baseline and 12 weeks]
  The difference of the mean of third and second recorded diastolic blood pressure readings on a seated relaxed patient from the battery powered digital blood pressure machine was recorded.
Mean's change from 12 weeks to 24 weeks in the seated patient through cuff mean diastolic blood pressure | [Time Frame: 12 weeks and 24 weeks]
  The difference of the means of third and second recorded diastolic blood pressure readings of the 12 and 24 weeks on a seated relaxed patient from the battery powered digital blood pressure machine was recorded.
Means' change from baseline in the seated patient through cuff mean diastolic blood pressure from 0 to 24 weeks | [Time Frame: baseline and 24 weeks]
  The difference of the means of third and second recorded systolic blood pressure readings of the 0 and 24 weeks on a seated relaxed patient from the battery powered digital blood pressure machine was recorded.
Means' change from baseline in the level of fasting blood sugar (mg/dl) | [Time-line: baseline, 12 weeks]
  Clinical chemistry laboratory test of blood sugar assesses using blood samples. The normal values are between 70 and 115 mg/dl. FBS≥ 115 = abnormal
Means change from 12 weeks in the level of fasting blood sugar (mg/dl) | [Time-line: 12 weeks, 24 weeks]
  Clinical chemistry laboratory test of blood sugar assessment using blood samples. The normal values are between 70 and 115 mg/dl. FBS≥ 115 = abnormal.
Means change from baseline in the level of fasting blood sugar (mg/dl) | [Time-line: 12 weeks, 24 weeks]
  Clinical chemistry laboratory test of blood sugar assessment using blood samples. The normal values are between 70 and 115 mg/dl. FBS≥ 115 = abnormal
Means change from baseline to 12 weeks in the level of total cholesterol (TC) (mg/dl) | [Time line: baseline, 12 weeks]
  Clinical chemistry laboratory test of lipids products assessment using blood sample. The normal value is values ≤ 200 mg/dl; beyond which you have hypercholesterolemia
Means change from 12 weeks to 24 in the level of total cholesterol (TC) (mg/dl) | [Time line: 12 weeks and 24 weeks]
  Clinical chemistry laboratory test of lipids products assessment using blood sample. The normal value is values ≤ 200 mg/dl; beyond which you have hypercholesterolemia
Means change from baseline to 24 weeks in the level of total cholesterol (TC) (mg/dl) | [Time line: baseline, 24 weeks]
  Clinical chemistry laboratory test of lipids products assessment using blood sample. The normal value is values < 200 mg/dl; beyond which you have hypercholesterolemia
Means change from baseline to 12 weeks in the level of High density lipoproteins (HDL) (mg /dl) | [Time line: baseline, 12 weeks]
  Change from baseline to 12 weeks in the level of high density lipoproteins (HDL) (mmol/dl) Clinical chemistry laboratory test of lipids products assessment using blood sample. The normal value is values ≤ >1.15 millimole per deciliter; beyond which you have high HDL
Means change from 12 weeks to 24 in the level of High density lipoproteins (HDL) (mg/dl) | [Time line: 12 weeks and 24 weeks]
  Clinical chemistry laboratory test of lipids products assessment using blood sample. The normal value is values ≤ 150 mg/dl; beyond which you have high HDL.
Means change from baseline to 24 weeks in the level of High density lipoproteins (HDL) (mg/dl) | [Time line: baseline, 24 weeks]
  Clinical chemistry laboratory test of lipids products assessment using blood sample. The normal value is values ≤ 150 mg/dl; beyond which you have high HDL
Means change from baseline to 12 weeks in the level of low density lipoproteins (LDL) (mg/dl) | [Time line: baseline, 12 weeks]
  Change from baseline to 12 weeks in the level of low density lipoproteins (LDL) (mg/dl) Clinical chemistry laboratory test of lipids products assessment using blood sample. The normal value is values ≤ 150 mg/dl; beyond which you have high LDL.
Means change from 12 weeks to 24 in the level of low density lipoproteins (LDL) (mg/dl) | [Time line: 12 weeks and 24 weeks]
  Clinical chemistry laboratory test of lipids products assessment using blood sample. The normal value is values ≤ 150 mg/dl; beyond which you have high LDL.
Means change from baseline to 24 weeks in the level of Low density lipoproteins (LDL) (mg/dl) | [Time line: baseline, 24 weeks]
  Clinical chemistry laboratory test of lipids products assessment using blood sample. The normal value is values ≤ 150 mg/dl; beyond which you have high LDL
Means change from baseline to 12 weeks in the level of triglycerides (TGC) (mg/dl) | [Time line: baseline, 12 weeks]
  Change from baseline to 12 weeks in the level of triglycerides (TGC) (mg/dl) Clinical chemistry laboratory test of lipids products assessment using blood sample. The normal value is values ≤ 203.5 mg/dl; beyond which you have high TGC
Means change from 12 weeks to 24 in the level of triglycerides (TGC) (mg/dl) | [Time line: 12 weeks and 24 weeks]
  Clinical chemistry laboratory test of lipids products assessment using blood sample. The normal value is values ≤ 203 mg/dl; beyond which you have high TGC
Means change from baseline to 24 weeks in the level of triglycerides (TGC) (mg/dl). | [Time line: baseline, 24 weeks]
  Clinical chemistry laboratory test of lipids products assessment using blood sample. The normal value is values ≤ 203.5 mg/dl; beyond which you have high TGC

CONTACTS AND LOCATIONS:
Overall Officials: Adamson S Muula, PhD, Study Director — Kamuzu University of Health Sciences
Locations (1):
- Mangochi District Hospital, Mangochi, Eastern-Region, Malawi

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: SAP, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: will to learn more or clarification on results will prompt to share IPD,all data data which may assist in clear understanding of the results. Once the request sent, it will be reviewed by the principal investigator. The criteria to review he request will be the seriousness of the request ( either in understanding the study or verification of the results, or will to reproduce the study within the ethical criteria regulations.

REFERENCES:
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] De Vet E, de Nooijer J, de Vries NK, Brug J. The Transtheoretical model for fruit, vegetable and fish consumption: associations between intakes, stages of change and stage transition determinants. Int J Behav Nutr Phys Act. 2006 Jun 19;3:13. doi: 10.1186/1479-5868-3-13. PMID 16784520
- [Background] Bush K, Kivlahan DR, McDonell MB, Fihn SD, Bradley KA. The AUDIT alcohol consumption questions (AUDIT-C): an effective brief screening test for problem drinking. Ambulatory Care Quality Improvement Project (ACQUIP). Alcohol Use Disorders Identification Test. Arch Intern Med. 1998 Sep 14;158(16):1789-95. doi: 10.1001/archinte.158.16.1789. PMID 9738608
- [Background] de Granda-Orive JI, Pascual-Lledo JF, Asensio-Sanchez S, Solano-Reina S, Garcia-Rueda M, Martinez-Muniz MA, Lazaro-Asegurado L, Bujulbasich D, Pendino R, Luhning S, Cienfuegos-Agustin I, Jimenez-Ruiz CA. Fagerstrom Test and Heaviness Smoking Index. Are they Interchangeable as a Dependence Test for Nicotine? Subst Use Misuse. 2020;55(2):200-208. doi: 10.1080/10826084.2019.1660680. Epub 2019 Sep 13. PMID 31519135
- [Background] Cleland C, Ferguson S, Ellis G, Hunter RF. Validity of the International Physical Activity Questionnaire (IPAQ) for assessing moderate-to-vigorous physical activity and sedentary behaviour of older adults in the United Kingdom. BMC Med Res Methodol. 2018 Dec 22;18(1):176. doi: 10.1186/s12874-018-0642-3. PMID 30577770
- [Background] Malan Z, Mash B, Everett-Murphy K. Evaluation of a training programme for primary care providers to offer brief behaviour change counselling on risk factors for non-communicable diseases in South Africa. Patient Educ Couns. 2016 Jan;99(1):125-31. doi: 10.1016/j.pec.2015.08.008. Epub 2015 Aug 14. PMID 26324109
- [Background] Amberbir A, Lin SH, Berman J, Muula A, Jacoby D, Wroe E, Maliwichi-Nyirenda C, Mwapasa V, Crampin A, Makwero M, Singogo E, Phiri S, Gordon S, Tobe SW, Masiye J, Newsome B, Hosseinipour M, Nyirenda MJ, van Oosterhout JJ. Systematic Review of Hypertension and Diabetes Burden, Risk Factors, and Interventions for Prevention and Control in Malawi: The NCD BRITE Consortium. Glob Heart. 2019 Jun;14(2):109-118. doi: 10.1016/j.gheart.2019.05.001. PMID 31324364
- [Background] Colbourn T, Masache G, Skordis-Worrall J. Development, reliability and validity of the Chichewa WHOQOL-BREF in adults in Lilongwe, Malawi. BMC Res Notes. 2012 Jul 3;5:346. doi: 10.1186/1756-0500-5-346. PMID 22759784
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- See also: book website used for training of health workers in brief behavior change counseling in South Africa . Which we adopted for our study. — https://www.ichange4health.co.za/wp-content/uploads/2016/01/HELPING-PEOPLE-CHANGE.pdf